CLINICAL TRIAL: NCT05880563
Title: A Monocentric, Controlled, Open Label, Phase I, First-in-human Trial to Investigate the Regional Distribution of [18F]RoSMA-18-d6 in the Brain and Spinal Cord to Assess Cannabinoid Type 2 Receptor (CB2R) Expression in Healthy Volunteers and Patients With Amyotrophic Lateral Sclerosis (ALS) by Positron Emission Tomography (PET)
Brief Title: Investigation of Cannabinoid 2-receptor Expression in the Brain and Spine of ALS-patients Compared to Healthy Controls With PET (18F-RoSMALS)
Acronym: 18F-RoSMALS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Markus Weber (Other)
Collaborators: ETH Zurich (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor-Investigator, Markus Weber, Prof. Dr. med., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18F-RoSMALS
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a controlled, open-label, first in man study to evaluate the regional distribution and brain-kinetics of [18F]RoSMA-18-d6 in ALS patients (n=20) and healthy volunteers (n=10).
  ALS patients will get two imaging sessions with [18F]RoSMA-18-d6 PET/CT and MRI-scans one year apart. Healthy volunteers will get only one pair of [18F]RoSMA-18-d6 PET/CT and MRI scans
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALS patients (Experimental): ALS patients will get two imaging sessions with [18F]RoSMA-18-d6 PET/CT and MRI-scans one year apart
  Interventions: Drug: [18F]-RoSMA-18-d6
- Healthy volunteers (Experimental): Healthy volunteers will get only one pair of [18F]RoSMA-18-d6 PET/CT and MRI scans
  Interventions: Drug: [18F]-RoSMA-18-d6

INTERVENTIONS:
Drug: [18F]-RoSMA-18-d6 — [18F]-RoSMA-18-d6 will be administered intravenously by a bolus injection followed by a subsequent PET/CT-scan of the brain and the spine

SUMMARY:
This clinical trial is a phase 1 study in which investigations with the weakly radioactive substance [18F]-RoSMA-18-d6 are being carried out for the first time.

This radiolabeled substance will be used to study a specific protein in the brain and spinal cord of patients with ALS and healthy individuals. This particular protein, the cannabinoid type 2 receptor, is thought to play a role in the disease process of ALS. Furthermore, it is assumed that this protein is found more frequently in the brain and spinal cord of patients with ALS compared to healthy individuals.

The following questions will be answered by this clinical trial.

1. Is this protein found, as suspected, increased in the brain and spinal cord of ALS patients compared to healthy individuals ?
2. Does the amount of this protein change during the course of the disease?
3. Are there any correlations between the observed changes in the amount of protein and the assessment of the course of the disease?

ELIGIBILITY:
Inclusion Criteria _ALS-patients:

* Age ≥18 years
* Able to provide written informed consent prior to study participation
* Body weight of ≥ 50 kg and a body mass index (BMI) between 19-30 kg/m2
* Vital signs measured after three minutes resting in the supine position must be within the following ranges:

  * oral body temperature: 35.0-37.5 °C
  * systolic blood pressure: 90-140 mm Hg
  * diastolic blood pressure: 50-90 mm Hg
  * pulse rate: 40-90 bpm
* Clinically probable, probable laboratory supported, or definite ALS-diagnosis according to the revised version of the El Escorial World Federation of Neurology criteria (EEC) (46)
* Disease duration ≤ 18 months since date of diagnosis
* Slow vital capacity (sVC) ≥ 80 % of normal (best of three measurements)
* Pre-study ALSFRS-R progression between disease onset and screening of -0.4 points/month or worse (calculated by ALSFRS-R score decline from 48 divided by months since symptom onset until screening)
* Patient has to be on a stable dose of disease modifying treatments (Edaravone 60 mg i.v.

on ten days/month, Riluzole 100 mg/day)

nclusion Criteria _Healthy controls

* Age ≥ 18 years
* Able to provide written informed consent prior to study participation
* Body weight of ≥ 50 kg and a body mass index (BMI) between 19-30 kg/m2
* Vital signs measured after 3 minutes resting in the supine position must be within the following ranges:

  * oral body temperature: 35.0-37.5 °C
  * systolic blood pressure: 90-140 mm Hg
  * diastolic blood pressure: 50-90 mm Hg
  * pulse rate: 40-90 bpm

Exclusion Criteria_ALS-patients

* Previous participation in another clinical study involving trial medication within the preceding 12 weeks prior to [18F]RoSMA-18-d6 administration
* Tracheostomy or continuous assisted ventilation of any type, or any other significant pulmonary disorder not attributed to ALS
* Structural brain or spinal cord abnormalities on MRI (e.g. evidence of stroke, infarct, or other space-occupying lesion or structural abnormality in brain and/or spinal cord.)
* Significant illness within two weeks prior to dosing
* History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug
* History of allergic reaction to drugs or anaphylactic shock.
* History of myocardial infarction or history of treated cancer[18F]RoSMA-18-d6 in ALS brain and spinal cord_ Version 1.1_29.11.2022 Page 45 of 98
* Current clinically significant systemic illness or symptoms (e.g., respiratory or cardiovascular disease) that may deteriorate or affect the patient's safety or ability to cooperate during the study.
* Gastrostomy
* Any medical condition known to have an association with motor neuron dysfunction or involving neuromuscular weakness or another neurodegenerative disease, e.g. Parkinson's Disease (PD) or Alzheimer's disease (AD), which might confound or obscure the diagnosis of ALS
* Major internal disorders (e.g. arterial hypertension, diabetes, evidence suggestive of liver or renal disease (bilirubin >1.6 mg/dL, creatinine > 150 μM).
* Presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment
* Donation or loss of 400 mL or more of blood within eight weeks prior to dosing.
* Clinically relevant abnormalities on blood screening (see 4.3.1)
* Use of any prescription drug with central action or over-the-counter (OTC) medication within two weeks prior to dosing, except ALS-medication and Paracetamol which are acceptable.
* Use of tobacco products in the previous three months
* History of drug (e.g. Cannabis) or alcohol abuse within 12 months prior to dosing
* Pregnancy or breast feeding

Exclusion criteria_healthy volunteers:

* Significant neurological or psychiatric disease
* Significant illness within two weeks prior to dosing
* History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug.
* History of myocardial infarction or history of treated cancer
* Current clinically significant systemic illness or symptoms (e.g., respiratory or cardiovascular disease) that may deteriorate or affect the patient's safety or ability to cooperate during the study.
* Major internal disorders (e.g. arterial hypertension, diabetes, evidence of suggestive liver or renal disease (bilirubin >1.6 mg/dL, creatinine > 150 μM).
* Other clinically significant abnormality on physical, neurological, or laboratory examination that, in the opinion of the investigator precludes the patient from the study.
* Clinically significant abnormality on electrocardiogram (ECG) that, in the opinion of the investigator, precludes the patient from the study.
* A past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome.
* Structural brain or spinal cord abnormalities on MRI (e.g., evidence of stroke, infarct, or other space-occupying lesion or structural abnormality in brain and/or spinal cord). History of allergic disease or anaphylactic shock.
* Presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment
* Use of any prescription drug or over-the-counter (OTC) medication within two weeks prior to dosing. Paracetamol is acceptable.
* Use of tobacco products in the previous three months.
* History of drug (e.g. Cannabis) or alcohol abuse within 12 months prior to dosing.
* Participation in any clinical investigation within four weeks prior to dosing or any ever participation in a research study with an amyloid lowering objective.
* Donation or loss of 400 mL or more of blood within eight weeks prior to dosing.
* Clinically relevant abnormalities on blood screening (see 4.3.1)
* Significant radiation exposure, especially in the last quarter (either X-ray or nuclear medicine studies). Any earlier nuclear medicine studies.
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Difference of [18F]RoSMA-18-d6 uptake in the brain and spinal cord between ALS patients (at baseline and day 360) and healthy, age- and gender-matched subjects, as assessed by PET and MRI to allow morphological mapping | Baseline and day 360
  Voxelwise maps of the total distribution volume (VT; ml g-
  1) of [18F]RoSMA-18-d6 are calculated using the Logan method (42) as well as compartmental modelling i.e., the evaluation of the microparameters of a two-tissue reversible binding model (43) Mean parametric maps for brain are calculated for the baseline and follow-up conditions in the controls and ALS patient groups. Furthermore, standardized uptake values (SUV) regarding tracer uptake after 15, 30, 60 and - if available - 90 minutes will be determined

SECONDARY OUTCOMES:
[18F]RoSMA-18-d6 uptake at month twelve (360 days) compared with uptake at baseline as assessed by PET/CT of the brain and spinal cord. | Baseline and day 360
Correlation of [18F]RoSMA-18-d6 uptake with corresponding ALSFRS-Score from baseline to day 360. | Baseline and day 360
Correlation of [18F]RoSMA-18-d6 uptake with corresponding respiratory function measurements (FVC, SNIP) from baseline to day 360. | Baseline and day 360
Correlation of the change of [18F]RoSMA-18-d6 endpoints (Δ-CB2R; baseline to day 360) with corresponding changes of the-ECAS score | Baseline and day 360

CONTACTS AND LOCATIONS:
Locations (1):
- Muskelzentrum/ALS-Clinic, Kantonsspital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No